CLINICAL TRIAL: NCT01538901
Title: Topical Imiquimod 5% Cream Therapy Versus Photodynamic Therapy With Methyl-aminolaevulinate 16% Cream of Actinic Keratoses in Organ Transplant Recipients
Brief Title: Imiquimod Versus Photodynamic Therapy of Actinic Keratoses in Organ Transplant Recipients
Acronym: AKtransplant
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: prolonged recruitment phase
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Stanislava Tzaneva, Doz. Dr., Medical University of Vienna
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPDTAKOTR/V06/28.12.11
Record Dates: First submitted 2012-02-19; First posted 2012-02-24 (Estimated); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Actinic Keratoses
Keywords: actinic keratoses; organ transplant recipients; photodynamic therapy; imiquimod
MeSH Terms: conditions — Keratosis, Actinic | interventions — Photochemotherapy; methyl 5-aminolevulinate; Imiquimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- photodynamic therapy (Experimental): Methyl-aminolaevulinate 16% cream (Metvix 160mg/g cream) will be applied 1 mm thick on the treated area, which has a maximal diameter of 8 cm2, and will be covered with a semipermeable dressing (Suprasorb F, Lohmann & Rauscher, Vienna, Austria)for 3 hours. Afterwards the cream leftovers will be removed by 0.9% NaCl solution. Following the treated area will be irradiated with heat-free visible red light at a peak wavelength of 630 nm with a single dose of 37 J/cm2 (Actilite model: CL128, PhotoCure, Norway). This treatment will be repeated in two weeks.
  Interventions: Other: photodynamic therapy
- imiquimod 5% cream (Active Comparator): 250 mg imiquimod 5% cream (Aldara 5% cream) will be applied over night, for a total of 3 nights in a week, for duration of 4 weeks.
  Interventions: Drug: imiquimod 5% cream

INTERVENTIONS:
Other: photodynamic therapy — Methyl-aminolaevulinate 16% cream (Metvix) will be applied on the treated area under occlusion for 3 hours. It follows irradiation with visible red light at a peak wavelength of 630 nm (Actilite CL128) with a single dose of 37 J/cm2.
  Other Names: Metvix 160mg/g cream photodynamic therapy
  Arms: photodynamic therapy
Drug: imiquimod 5% cream — 250 mg imiquimod 5% cream will be applied over night for a total of 3 nights in the week, for duration of 4 weeks
  Other Names: Aldara 5% cream
  Arms: imiquimod 5% cream

SUMMARY:
The purpose of this study is to compare two different therapies for actinic keratoses in organ transplant recipients with regard to efficacy and tolerability. The investiagtors are planning to examine treatment with Imiquimod 5% cream versus treatment with Methyl-aminolaevulinate 16% cream and subsequent irradiation with red light, so-called photodynamic therapy, in this patients' group. A secondary objective of our study is to investigate the reduction in the field cancerisation after both treatments using fluorescence diagnostic method and digital imaging.

DETAILED DESCRIPTION:
Organ transplant patients (OTP) require lifelong immunosuppressive therapy and consequently are prone to develop skin tumors, i.e skin cancer is the most frequent malignancy in organ transplant recipients. OTP frequently develop extensive areas of actinic damage, epidermal dysplasia, wich accounts for increased risk of aggressive skin cancer development in susceptible patients, and are referred to as "field cancerisation". Therefore the whole area of field cancerisation has to be treated. In our study we will treat this areas with two different methods and not only the single visible lesions of actinic keratoses.In this open prospective randomized intraindividual study one half of the patients' scalp or face will be treated with Imiquimod 5% cream for 4 weeks, 3 times a week, and the other half with Methyl-aminolaevulinate 16% cream photodynamic therapy, two applications in two weeks interval. The pre- and post treatment extension of field cancerisation will be assessed by means of a highly sensitive digital fluorescence imaging system.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Patients who had received a kidney, liver, lung or heart transplant more than 3 years prior to inclusion into the study
* Patients who had been treated at least 6 months prior to study entry with a stable twofold or threefold immunosuppressive treatment
* Patients who had clinically confirmed epithelial dysplasia (actinic keratoses) in at least two anatomically separated contralateral areas on the face and/or scalp with comparable size and extension and minimum distance of 5 cm

Exclusion Criteria:

* Invasive squamous cell carcinoma or basal cell carcinoma in the treatment area
* Known allergy to imiquimod and/or methyl-aminolaevulinate and/or one of the other components of the investigational products and/or peanut oil
* Patients who have received retinoids, interferons or investigational drugs within 4 weeks of study initiation
* Patients who are participating in othe dermatological study
* Persistent Hepatitis B or C infections
* Any evidence of systemic cancer
* Patients who have received any systemic cancer chemotherapy or radiation therapy
* Pregnant or lactating women
* Patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Clinical complete response rate of actinic keratoses | 4 weeks after end of treatment
  The clinical complete response rate of actinic keratoses is defined as a proportion of the number of actinic keratoses with a clinically determined complete clearance(no visible and/or palpable actinic keratoses) to the number of the actinic keratoses at baseline.

SECONDARY OUTCOMES:
clinical complete response rate of actinic keratoses | 6 and 12 months after end of treatment
  The clinical complete response rate of actinic keratoses is defined as a proportion of the number of actinic keratoses with a clinically determined complete clearance(no visible and/or palpable actinic keratoses) to the number of the actinic keratoses at baseline.
global reduction in the area of specific fluorescence | 1, 6 and 12 months after end of treatment
  Prior to photodynamic therapy an illumination of the treated area with a Wood light will be prepared (fluorescence diagnostik). The specific fluorescence will be detected and documented using the non-invasive fluorescence-imaging system Dyaderm, Biocam, Germany.
global patient's satisfaction | 3, 6 and 12 months after end of treatment
  The global patient's satisfaction will be determined by the patients themselves on a 10 cm visual analog scale. 0 means extremely unsatisfied, 1-3 means unsatisfied, 5-7 means moderately satisfied, 8-10 means highly satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Stanislava Tzaneva, Doz. Dr., Principal Investigator — Medical University of Vienna, University Clinic of Dermatology, Division of General Dermatology; Alexandra Geusau, Prof. Dr., Principal Investigator — Medical University of Vienna, Division of Immunology, Allergy and Infectious Diseases
Locations (2):
- Austria (2):
  - Medical University of Vienna, University Clinic of Dermatology, Vienna
  - Medical University of Vienna, Vienna

REFERENCES:
- [Background] Ulrich C, Bichel J, Euvrard S, Guidi B, Proby CM, van de Kerkhof PC, Amerio P, Ronnevig J, Slade HB, Stockfleth E. Topical immunomodulation under systemic immunosuppression: results of a multicentre, randomized, placebo-controlled safety and efficacy study of imiquimod 5% cream for the treatment of actinic keratoses in kidney, heart, and liver transplant patients. Br J Dermatol. 2007 Dec;157 Suppl 2(Suppl 2):25-31. doi: 10.1111/j.1365-2133.2007.08269.x. PMID 18067628
- [Background] Dragieva G, Prinz BM, Hafner J, Dummer R, Burg G, Binswanger U, Kempf W. A randomized controlled clinical trial of topical photodynamic therapy with methyl aminolaevulinate in the treatment of actinic keratoses in transplant recipients. Br J Dermatol. 2004 Jul;151(1):196-200. doi: 10.1111/j.1365-2133.2004.06054.x. PMID 15270891
- [Background] Stockfleth E, Ulrich C, Meyer T, Christophers E. Epithelial malignancies in organ transplant patients: clinical presentation and new methods of treatment. Recent Results Cancer Res. 2002;160:251-8. doi: 10.1007/978-3-642-59410-6_30. PMID 12079221
- [Background] Stern RS, Bolshakov S, Nataraj AJ, Ananthaswamy HN. p53 mutation in nonmelanoma skin cancers occurring in psoralen ultraviolet a-treated patients: evidence for heterogeneity and field cancerization. J Invest Dermatol. 2002 Aug;119(2):522-6. doi: 10.1046/j.1523-1747.2002.01814.x. PMID 12190879
- [Background] Geusau A, Dunkler D, Messeritsch E, Sandor N, Heidler G, Rodler S, Ankersmit J, Zuckermann A, Tschachler E. Non-melanoma skin cancer and its risk factors in an Austrian population of heart transplant recipients receiving induction therapy. Int J Dermatol. 2008 Sep;47(9):918-25. doi: 10.1111/j.1365-4632.2008.03711.x. PMID 18937654
- [Background] Fernandez-Guarino M, Harto A, Sanchez-Ronco M, Perez-Garcia B, Marquet A, Jaen P. [Retrospective, descriptive, observational study of treatment of multiple actinic keratoses with topical methyl aminolevulinate and red light: results in clinical practice and correlation with fluorescence imaging]. Actas Dermosifiliogr. 2008 Dec;99(10):779-87. Spanish. PMID 19091216